CLINICAL TRIAL: NCT06427317
Title: Routinely Collected Clinical Data and Evaluation of Antimicrobial Target Attainment and the Potential Role of Therapeutic Drug Monitoring in UK Infection Management
Brief Title: Routinely Collected Clinical Data and Evaluation of Antimicrobial Target Attainment
Acronym: DATATDM
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 21HH7287
Record Dates: First submitted 2024-03-27; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Infections, Bacterial; Pharmacokinetics; Drug Monitoring; Drug-Related Side Effects and Adverse Reactions
MeSH Terms: conditions — Bacterial Infections; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sera, saliva, urine, nasal mucous, CSF, renal replacement fluid, CSF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary aim of the study is to determine the proportion of individuals receiving beta-lactam antibiotics at Imperial College Healthcare NHS Trust in whom drug concentration targets are achieved.

DETAILED DESCRIPTION:
To address the challenge of antimicrobial resistance (AMR) it is imperative that the current finite pool of antimicrobial agents is optimised, to maximise therapeutic success, limit the risk of drug toxicity, whilst minimising emergence of resistance.

Outside of the critical care setting it is not known how many patients are receiving optimal drug concentrations for the treatment of infection.

This study aims to assess whether antimicrobial targets are being achieved in these individuals and explore how clinical co-variates and outcomes may relate to this. Furthermore, it aims to identify priority groups and/or drugs where there are gaps in dose optimisation research and develop hypotheses which can be tested in observational studies.

Eligible participants will be enrolled and observed during their management of infection at Imperial College NHS Trust. After providing informed consent their clinical data will be collected from electronic healthcare records and they will provide samples that will undergo drug concentration analysis.

ELIGIBILITY:
Inclusion Criteria:

18 years of age or above.

* Under follow-up for management of infection at Imperial College NHS Trust
* Received a beta-lactam antibiotic within the last 48 hours (or are planned to start imminently).
* Provides informed written consent see below, or lacks capacity to provide consent because of one of the following conditions (and declaration provided by personal consultee):
* Delirium which may be caused or exacerbated by having an infection.
* Suspected/confirmed central nervous system infection.
* Critical illness requiring sedation and/or intubation and ventilation which is caused by or exacerbated by having an infection.

Exclusion Criteria:

* Less than 18 years of age

  * Severe anaemia (Hb < 70g/l)
  * Platelets < 50x10^9/l, INR >1.5 or other known blood clotting impairment
  * Patient with terminal diagnosis receiving palliative care input who may experience distress if approached for this study.
  * Enrolled in a clinical trial which stipulates exclusion from other studies including observational studies.
  * Patients with restricted liberty, prisoners or under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As per inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 323 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2027-03-19 (Estimated); Study Completion 2027-03-19 (Estimated)

PRIMARY OUTCOMES:
Determine the number of individuals receiving beta-lactam antibiotics at Imperial College Healthcare NHS Trust in whom drug concentration targets are achieved. | 3 years
  Determine the number of individuals receiving beta-lactam antibiotics at Imperial College Healthcare NHS Trust in whom drug concentration targets are achieved

SECONDARY OUTCOMES:
Find the number of individuals receiving co-administered non-beta-lactam antibiotics in whom drug concentration targets are achieved. | 3 years
  Find the number of individuals receiving co-administered non-beta-lactam antibiotics in whom drug concentration targets are achieved.
Show how clinical co-variates, co-administered medications and treatment outcomes relate to target attainment, and identify groups of patients in who therapeutic drug monitoring may be beneficial. | 3 years
  Show how clinical co-variates, co-administered medications and treatment outcomes relate to target attainment, and identify groups of patients in who therapeutic drug monitoring may be beneficial.
Illustrate dynamic patterns of infection-related biomarkers which may indicate the presence/absence of treatment response. | 3 years
  Illustrate dynamic patterns of infection-related biomarkers which may indicate the presence/absence of treatment response.
Show how drug-levels obtained through minimally invasive sampling and the use of residual specimens relate to blood, and how these could be used to inform individual dose-optimisation. | 3 years
  Show how drug-levels obtained through minimally invasive sampling and the use of residual specimens relate to blood, and how these could be used to inform individual dose-optimisation.
Build a repository of real life PK-PD data which can be used to generate hypotheses and guide the development of interventional dose optimisation studies | 3 years
  Build a repository of real life PK-PD data which can be used to generate hypotheses and guide the development of interventional dose optimisation studies

CONTACTS AND LOCATIONS:
Overall Officials: Alison Holmes, MD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided